CLINICAL TRIAL: NCT05116176
Title: TRAjectories and CLinical ExpeRiences of ICD Therapy Study
Acronym: TRACER-ICD
Status: Enrolling by invitation | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Pennsylvania (Other); Hebrew SeniorLife (Other); University of Colorado, Denver (Other); Emory University (Other); Mayo Clinic (Other); Saint Luke's Health System (Other)
Responsible Party: Principal Investigator, Daniel B. Kramer, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2021P000054
Record Dates: First submitted 2021-03-12; First posted 2021-11-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Implantable Defibrillator User
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Implantable cardioverter-defibrillators — 500 patients age >65 receiving new primary prevention implantable cardioverter-defibrillators (ICDs).

SUMMARY:
This is a prospective cohort study of older patients receiving implantable cardioverter-defibrillators. The purpose of the TRACER-ICD study is to conduct a prospective cohort investigation with the goal of 500 patients age >65 receiving new primary prevention implantable cardioverter-defibrillators (ICDs). Patients will be followed quarterly for 18 months with interviews, electronic record review, and remote monitoring to characterize clinical and functional trajectories following device implantation, with permission for extended electronic follow-up for up to 10 years (Aim 1). This cohort will support validation and refinement of an established model for predicting personalized outcome profiles for ICD therapies and death (Aim 2). Lastly, we will combine electronic record review with semi-structured interviews with patients and physicians to evaluate physician and patient experiences with a prototype individualized shared decision-making (SDM) tool (Aim 3).

DETAILED DESCRIPTION:
Study Objectives and Design

The specific aims, applicable methods, and main hypotheses of the TRACER-ICD study are as follows:

Aim 1: To characterize the clinical course of patients aged >65 after ICD implantation by establishing a multicenter prospective cohort (N=500). Baseline (verbal and in-person) and quarterly (phone, electronic health records [EHR], remote monitoring) data collected up to 18 months or death will include: a. geriatric assessments (e.g. frailty, cognition,1 functional status; b. comorbidities; c. quality of life and symptom burden; d. health services use; e. SDM history; and f. ICD-recorded physical activity (minutes/day).

Factors associated with death and poor quality of life will be identified. Group-based trajectory modeling will identify patient clusters with distinct trajectories of functional status and quality of life following ICD implantation.

H1: A model integrating frailty and clinical factors will predict (a) death, (b) poor quality of life, and (c) unfavorable functional trajectories after ICD implantation.

Aim 2: To validate a personalized prediction model of treatment outcomes of ICDs. We will apply our established semi-competing risks approach5 to the prospective cohort, enriched by the baseline geriatric assessments, to predict individual patients' probabilities of the following outcome profiles at 6, 12, and 18 months post-implant: a. death without prior shock, b. death with prior shock, c. survival without prior shock, and d. survival with prior shock. The independent contribution of frailty, cognitive dysfunction, baseline quality of life, and functional status (e.g. total deficits in ADL and IADL) to model performance will be evaluated.

H2: Addition of frailty, cognitive dysfunction, quality of life, and functional status to a model with cardiovascular variables will significantly improve model performance as assessed by area under the curve (AUC).

Aim 3: To identify optimal strategies for incorporating personalized outcome profiles into SDM. The main cohort's baseline interview and EHR review will provide quantitative data on past SDM tools used by physicians. We will develop a prototype individualized version of the Colorado SDM tool that incorporates 18-month outcome profiles using our semi-competing risk model. We will perform semi-structured interviews of cardiologists (N=20) as well as patients (N=20) recruited from the main cohort regarding process mapping of SDM from clinic to implant procedure, including timing, content, format preferences, and impressions of the prototype individualized tool.

ELIGIBILITY:
Patients scheduled for ICD implantation will be identified at participating sites by site staff. Eligibility criteria will include the following, all of which must be met by all participants for participation:

1. Patient receiving new primary prevention ICD (single, dual chamber, or subcutaneous system)
2. Age >65 years
3. English-speaking (assessment instruments are only available/validated in English)
4. Sufficient cognitive ability to provide consent (i.e. answer simple questions on study participation, purpose and procedures)

Candidates meeting the following exclusion criteria at baseline will be excluded from study participation:

1. Receipt of cardiac resynchronization therapy device
2. Participation in another investigational drug or intervention trial expected to influence any of the outcomes of interest in this study
3. Current drug or alcohol use or dependence that, in the opinion of the Site Principle Investigator, would interfere with adherence to study requirements.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients scheduled for ICD implantation will be identified at participating sites by site staff. Eligibility criteria will include the following, all of which must be met by all participants for participation:
  1. Patient receiving new primary prevention ICD (single, dual chamber, or subcutaneous system)
  2. Age >65 years
  3. English-speaking (N.B.: assessment instruments are only available/validated in English)
  4. Sufficient cognitive ability to provide consent (i.e. answer simple questions on study participation, purpose and procedures)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Trajectories after ICD implantation | Patients will be followed quarterly for 18 months or to death.
  Group-based trajectory modeling will identify patient clusters with distinct trajectories of functional status and quality of life following ICD implantation.
Outcomes after ICD Implantation | Up to 18 months
  Death/Poor Quality of Life (combined endpoint)
Semi-competing risks model of deaths and/or ICD shocks | Up to 18 months
  Personalized outcome profiles for death +/- ICD shocks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Kramer, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No